CLINICAL TRIAL: NCT04187573
Title: Coil Assisted Flow Diversion: A Prospective, Single Arm, Multi-center Study to Assess the Safety and Performance of Neqstent in Adjunctive Therapy (CAFI Study)
Brief Title: Coil Assisted Flow Diversion Safety and Performance Study
Acronym: CAFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerus Endovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNQS428-01
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, multi-center study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Neqstent — Adjunctive device providing stable aneurysm neck coverage for the placement of embolization coils within the aneurysm sac and long term stable occlusion of the aneurysm.

SUMMARY:
Cerus Endovascular is sponsoring a prospective, single arm, multi-center study to document the safety and performance of Neqstent in adjunctive therapy.

The purpose of the study is to document safety and performance of the Neqstent in adjunctive therapy in treatment for patients with intracranial aneurysms (IA).

DETAILED DESCRIPTION:
Neqstent is designed as an adjunctive therapy for patients with unruptured and failed bifurcation aneurysm embolizations. Neqstent can be positioned at the neck of the aneurysm with or without existing coils and other embolization products. Embolization coils should be added to fill the dome of the aneurysm after placement of Neqstent.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's indication for treatment of unruptured IAs according to the national/international guidelines.
2. Age 18-80 years at screening
3. Patients who are suitable for non-emergency endovascular embolization of saccular IAs
4. IA located at a bifurcation in the anterior or posterior circulation with dimensions consistent with implant size selection guidelines included in the IFU
5. Patient has the necessary mental capacity to participate and is willing and able to participate in the study for the duration of the study follow-up and is able to comply with study requirements
6. Patient able to able to give their informed consent can be included in this study. This must be demonstrated by means of a personally signed and dated informed consent document indicating that the subject has been informed of and understood all pertinent aspects of the study.

Exclusion Criteria:

1. Ruptured aneurysm
2. Patient anatomy or physiology considered unsuitable for endovascular treatment
3. Any patient anatomy, physiology, existing implants with failed aneurysm embolization that would interfere with the ability for Neqstent to seal at the neck of the aneurysm. (i.e., compacted coils in close proximity to the neck that prevent good apposition of the Neqstent to the wall of the aneurysm, stent and/or stent-like devices whose struts span the aneurysm neck to retain the coil mass that inhibit access and/or successful Neqstent seating at the aneurysm neck, and/or any aneurysm that has a failed device and confirmed thrombus-burden inside the aneurysm sac)
4. Contraindication for arterial access
5. Largest measured IA neck diameter >8 mm or <3 mm
6. Target IA contains other devices/implants (e.g., coils) that will prevent complete expansion of Neqstent
7. Known allergy to platinum, nickel or titanium
8. Known allergy to contrast agents
9. Contraindication to anticoagulants or platelet inhibitor medication
10. Stenosis of the target IA's parent vessel >50%
11. Anticoagulation medications such as warfarin that cannot be discontinued.
12. Pregnant, breastfeeding or women of childbearing potential not on adequate birth control (only women with a highly effective method of contraception [oral contraception or intra-uterine device] or sterile women can be enrolled to the study)
13. Acute / chronic renal failure (including dialysis); Creatinine > 2.00 mg/dl or > 182 μmol/L
14. Myocardial Infarction, Stroke or TIA within the last 6 months
15. Any other medical issue within the brain that precludes the device implantation such as brain surgery, radiation in the target area of intervention, acute traumatic craniocerebral injury, etc.
16. Other medical conditions that cause an inability to comply with study requirements and/or that could increase the risk of neurovascular procedures or death within 2 years (e.g., liver failure, cancer, heart failure, chronic obstructive pulmonary disease, immunosuppression, neural disease, and hematologic disorders etc.)
17. Participating in another study with investigational devices or drugs that would confound the effects of the study outcomes
18. The presence of condition that may create unacceptable risk during the aneurysm embolization procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Liebig, MD, Principal Investigator — Klinikum der Universität München
Locations (7):
- Christian Doppler Klinikum, Salzburg, Austria
- Alberta Health Sciences, Edmonton, Alberta, Canada
- Odense University Hospital, Odense, Denmark
- Germany (3):
  - UK Hamburg, Hamburg
  - UKSH Kiel, Kiel
  - Klinikum der Universität München, Munich
- Inerespital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liebig T, Gal G, O Kelly C, Wodarg F, Killer-Oberpfalzer M, Ozpeynirci Y, Bester M, Tsogkas I, Psychogios MN, Jansen O, Fiehler J. Neqstent coil-assisted flow diverter (NQS) for the treatment of bifurcation aneurysms: the coil-assisted flow diversion safety and performance study (CAFI). J Neurointerv Surg. 2024 Jun 17;16(7):721-725. doi: 10.1136/jnis-2022-020056. PMID 37419693
- See also: Sponsor Web-site — http://cerusendo.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention/Neqstent: Device: Neqstent Adjunctive device providing stable aneurysm neck coverage for the placement of embolization coils within the aneurysm sac and long term stable occlusion of the aneurysm.
Period: Overall Study
Arm/Group | Intervention/Neqstent
Started | 38
Completed | 32
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: All patients; 38 patients were listed in the Participant Flow, and all 38 patients were included in the population description.
Arm/Group | Intervention/Neqstent
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5
  Austria | 2
  Denmark | 17
  Switzerland | 1
  Germany | 13

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With Death of Any Non-accidental Cause or Any Major Disabling Stroke After Treatment or Major Disabling Stroke or Death Due to Neurological Cause.
Time Frame: From day 31 to 6 months after treatment
Population: Intent-to-treat: All eligible subjects who underwent an attempt with the Neqstent device
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention/Neqstent
Number analyzed (Participants) | 37
Participants | 2

2. Primary Outcome: The Proportion of Subjects With Complete Occlusion
Description: Success will be defined as complete occlusion demonstrated by a Grade 1 using the Raymond Roy Scale.
Time Frame: 6 months
Population: Intent-to-treat: All eligible subjects who underwent an attempt with the Neqstent device.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention/Neqstent
Number analyzed (Participants) | 32
Participants | 26

ADVERSE EVENTS:
Time Frame: 2 years
Description: Per protocol, the SAE definition includes adverse events where medical or surgical intervention was necessitated to prevent life-threatening illness.
  Note: Planned hospitalization for a pre-existing condition, or a procedure required by the clinical investigational plan, without serious deterioration in health, is not considered to be an SAE.
Arm/Group | Intervention/Neqstent
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 15/37
Other Adverse Events (participants affected / at risk) | 19/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention/Neqstent (N=37)
Aneurysm Reccurence (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 7 (9)
Headache (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Shoulder Injury (Injury, poisoning and procedural complications) | 1 (1)
Distal Embolic Phenomenon (Nervous system disorders) | 1 (1)
Hemorrhagic Stroke (Nervous system disorders) | 1 (1)
Device Movement (Investigations) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Target Aneurysm Rupture (Injury, poisoning and procedural complications) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Access Site - Hematoma (Vascular disorders) | 1 (1)
Non-index Aneurysm Treatment (Nervous system disorders) | 2 (2)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention/Neqstent (N=37)
Access Site - Hematoma (Vascular disorders) | 4 (4)
Headache and Nosebleed (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Stroke (Nervous system disorders) | 1 (1)
Disorientation with trouble speaking (General disorders) | 1 (1)
Tinnitus (Nervous system disorders) | 1 (1)
Dental Surgery (Surgical and medical procedures) | 1 (1)
Radiation induced epilation (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)
Femoral Artery Dissection (Injury, poisoning and procedural complications) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
Vasovagal Episode (Cardiac disorders) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1)
Fractured Fibula (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary Abcess (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bleeding Event (Non-neurological) (General disorders) | 1 (1)
Dizziness/Fall (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT04187573/Prot_SAP_000.pdf